CLINICAL TRIAL: NCT02901951
Title: Long-term Persistence of Immunity to Hepatitis B in Adults Vaccinated 20 to 30 Years Ago With Engerix-B
Brief Title: Long-term Persistence of Immunity to Hepatitis B in Adults Vaccinated With GlaxoSmithKline (GSK) Biologicals' Hepatitis B Vaccine (HBV), Engerix-B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116811; 2015-004099-31 (EudraCT Number)
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B surface antigen antibody; adult subjects; Hepatitis B; HBV
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B

ARMS (1):
- HBV Group (Experimental): Subjects aged 40 to 60 years old who received 3 or 4 doses of Engerix-B (HBV vaccine) 20 to 30 years ago and were administered with a single challenge dose of HBV vaccine in this study at Day 0 (Visit 1).
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: Engerix-B — Intramuscular administration of single challenge dose of Engerix-B vaccine in the deltoid region of the non-dominant arm.

SUMMARY:
The purpose of this study is to assess the long-term protection against HBV infection in adult subjects, aged 18-40 years vaccinated with three or four doses of Engerix-B 20 to 30 years ago

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between and including 40 and 60 years of age (from and including the 40th birthday up to, but excluding, the 61st birthday) at the time of the vaccination.
* Written informed consent obtained from the subject.
* Documented evidence of previous vaccination with three or four consecutive doses of Engerix-B administered in adulthood (i.e. at least 18 years of age) with

  * the last dose received 4 to 12 months after the previous one,
  * no subsequent booster dose ever received later, and
  * the last dose received 20 to 30 years before enrolment.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for one month after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Previous hepatitis B booster vaccination since completion of the primary vaccination series with three or four doses of Engerix-B.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days preceding the dose of study vaccine, or planned administration during the study period, with the exception of seasonal influenza vaccine.
* Any medical condition that in the judgment of the investigator places the subject at undue risk by participating in the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* History of hepatitis B disease or episode of jaundice with unknown etiology.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Major congenital defects or serious chronic illness (including insulin-dependent diabetes).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C for oral, axillary or tympanic route, or 38.0°C on rectal route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the dose of study vaccine, or planned administration during the study period.
* Drug and/ or alcohol abuse within the last 5 years.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Wilrijk
- Canada (2):
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=116811

REFERENCES:
- [Background] Van Damme P, Dionne M, Leroux-Roels G, Van Der Meeren O, Di Paolo E, Salaun B, Surya Kiran P, Folschweiller N. Persistence of HBsAg-specific antibodies and immune memory two to three decades after hepatitis B vaccination in adults. J Viral Hepat. 2019 Sep;26(9):1066-1075. doi: 10.1111/jvh.13125. Epub 2019 Jun 2. PMID 31087382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects aged between and including 40 to 60 years were enrolled in this study, in compliance with the inclusion criteria, which required the documented evidence of previous vaccination with three or four consecutive doses of Engerix-B administered in adulthood (i.e. at least 18 years of age).
Pre-assignment Details: 106 subjects were enrolled in the study but 3 subjects were withdrawn before vaccine administration. Therefore, the number of subjects started is 103.
Period: Overall Study
Arm/Group | HBV Group
Started | 103
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HBV Group: Subjects aged 40 to 60 years old who received 3 or 4 doses of HBV vaccine 20 to 30 years ago and were administered with a single challenge dose of HBV vaccine in this study at Day 0 (Visit 1).
Arm/Group | HBV Group
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With an Anamnestic Response to the HBV Challenge Dose, Based on the Last Available Time Point Before the Challenge Dose
Description: Anamnestic response to the challenge dose was defined as: At least (i.e. greater than or equal to [≥]) 4-fold rise in one month post-vaccination anti-hepatitis B surface antigen (anti-HBs) antibody concentrations in previously seropositive subjects (Subjects with anti-HBs antibody concentration ≥ 6.2 milli International Unit/Milliliter (mIU/mL) at the pre-challenge dose time point); In previously seronegative subjects (Subjects with anti-HBs antibody concentration < 6.2 mIU/mL at the pre-challenge dose time point), anti-HBs antibody concentrations ≥10 mIU/mL at one month post-challenge dose time-point.
Time Frame: 7 days after the challenge dose (Day 7)
Population: Analysis was performed on the According-to-protocol (ATP) cohort for analysis of immunogenicity which included all evaluable subjects who had received the challenge dose of HRV vaccine and for whom data concerning immunogenicity outcome measures at pre-challenge (Day 0) and one month post-challenge (Day 30) were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HBV Group
Number analyzed (Participants) | 101
Percentage of subjects
  < 6.2 mIU/mL: number analyzed (Participants) | 6
  < 6.2 mIU/mL | 66.7 [22.3 to 95.7]
  ≥ 6.2 mIU/mL: number analyzed (Participants) | 95
  ≥ 6.2 mIU/mL | 85.3 [76.5 to 91.7]

2. Primary Outcome: Percentage of Subjects With an Anamnestic Response to the HBV Challenge Dose, Based on the Last Available Time Point Before the Challenge Dose
Description: Anamnestic response to the challenge dose was defined as: At least (i.e. ≥ 4-fold rise in one month post-vaccination anti-HBs antibody concentrations in previously seropositive subjects (Subjects with anti-HBs antibody concentration ≥ 6.2 mIU/mL at the pre-challenge dose time point); In previously seronegative subjects (Subjects with anti-HBs antibody concentration < 6.2 mIU/mL at the pre-challenge dose time point), anti-HBs antibody concentrations ≥10 mIU/mL at one month post-challenge dose time-point.
Time Frame: 30 days after the challenge dose (Day 30)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity which included all evaluable subjects who had received the challenge dose of HRV vaccine and for whom data concerning immunogenicity outcome measures at pre-challenge (Day 0) and one month post-challenge (Day 30) were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HBV Group
Number analyzed (Participants) | 101
Percentage of subjects
  < 6.2 mIU/mL: number analyzed (Participants) | 6
  < 6.2 mIU/mL | 100 [54.1 to 100]
  ≥ 6.2 mIU/mL: number analyzed (Participants) | 95
  ≥ 6.2 mIU/mL | 100 [96.2 to 100]

3. Secondary Outcome: Percentage of Subjects With Anti-HBs Antibody Concentrations Equal to or Above Cut-off Values
Description: Percentage of subjects with anti-HBs antibody concentrations ≥ 6.2 mIU/mL, ≥ 10 mIU/mL and ≥ 100 mIU/mL.
Time Frame: At the pre-challenge dose time-point (Day 0), at 7 days post-challenge time-point (Day 7) and at 30 days post-challenge time-point (Day 30)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | HBV Group
Number analyzed (Participants) | 101
Percentage of subjects
  ≥ 6.2 mIU/mL [Day 0] | 94.1 [87.5 to 97.8]
  ≥ 10 mIU/mL [Day 0] | 90.1 [82.5 to 95.1]
  ≥ 100 mIU/mL [Day 0] | 61.4 [51.2 to 70.9]
  ≥ 6.2 mIU/mL [Day 7] | 98.0 [93.0 to 99.8]
  ≥ 10 mIU/mL [Day 7] | 97.0 [91.6 to 99.4]
  ≥ 100 mIU/mL [Day 7] | 92.1 [85.0 to 96.5]
  ≥ 6.2 mIU/mL [Day 30] | 100 [96.4 to 100]
  ≥ 10 mIU/mL [Day 30] | 100 [96.4 to 100]
  ≥ 100 mIU/mL [Day 30] | 98.0 [93.0 to 99.8]

4. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Anti-HBs antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL.
Time Frame: At the pre-challenge dose time-point (Day 0), at 7 days post-challenge dose time-point (Day 7) and at 30 days post-challenge dose time-point (Day 30)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBV Group
Number analyzed (Participants) | 101
mIU/mL
  At Day 0 | 184.6 [121.5 to 280.3]
  At Day 7 | 3840.0 [2330.0 to 6328.6]
  At Day 30 | 48999.1 [33572.7 to 71513.7]

5. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Assessed solicited local symptoms were injection site pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after the challenge dose
Population: Analysis was performed on the Total Vaccinated cohort (TVC) which included all subjects who received the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 103
Participants
  Any Pain | 40
  Any Redness (mm) | 4
  Any Swelling (mm) | 3

6. Secondary Outcome: Number of Subjects With Any Solicited General AEs
Description: Assessed solicited general symptoms were fatigue, fever (defined as axillary temperature ≥ 37.5 degrees Celsius [°C]) , gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain) and headache. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after the challenge dose
Population: Analysis was performed on the TVC which included all subjects who received the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 103
Participants
  Any Fatigue | 27
  Any Gastrointestinal symptoms | 10
  Any Headache | 20
  Any Fever | 0

7. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after the challenge dose
Population: Analysis was performed on the TVC which included all subjects who received the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 103
Participants | 41

8. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed included any untoward medical occurrences that resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or congenital anomaly/birth defect in the offspring of a study subject. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Day 0 to Day 30)
Population: Analysis was performed on the TVC which included all subjects who received the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | HBV Group
Number analyzed (Participants) | 103
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited local & general AEs: during 4-day (Days 0-3) follow-up period after challenge dose; Unsolicited AEs: during 31-day (Days 0-30) follow-up period after challenge dose; SAEs: during the entire study period (Day 0 to Day 30).
Arm/Group | HBV Group
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 75/103
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBV Group (N=103)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Eye pruritus (Eye disorders) | 2 (2)
Fatigue (General disorders) | 29 (30)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (10)
Headache (Nervous system disorders) | 25 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Injection site erythema (General disorders) | 4 (4)
Injection site pain (General disorders) | 40 (40)
Injection site pruritus (General disorders) | 1 (1)
Injection site swelling (General disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Pyrexia (General disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT02901951/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02901951/SAP_001.pdf